CLINICAL TRIAL: NCT02760355
Title: Hepatitis C Virus Infection Induced Insulin Resistance: Different Contribution From Liver and Extrahepatic Sites as Inferred by Treating Chronic Hepatitis C Patients With an Interferon-free Antiviral Combination
Brief Title: Extrahepatic Insulin Resistance in Chronic Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Gastaldi Giacomo (Unknown); Clément Sophie (Unknown)
Responsible Party: Principal Investigator, Negro Francesco, Professor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-063
Record Dates: First submitted 2016-04-30; First posted 2016-05-03 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — ledipasvir; Sofosbuvir; ledipasvir, sofosbuvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active treatment (Experimental): Ledipasvir 90 mg/Sofosbuvir 400 mg, one tablet once a day + b.w. dose adjusted, 200 mg-tablets of ribavirin (1,000 mg in two administration in patients <75 Kg of body weight, or 1,200 mg in two administrations for those >75 Kg) for 12 weeks
  Interventions: Drug: Ledipasvir 90 mg/Sofosbuvir 400 mg; Drug: Ribavirin

INTERVENTIONS:
Drug: Ledipasvir 90 mg/Sofosbuvir 400 mg — Oral administration on one fixed dose combination tablet for 12 weeks
  Other Names: Harvoni
Drug: Ribavirin — Oral administration of body weight-dose adjusted, 200 mg-tablets of ribavirin (1,000 mg in two administration in patients <75 Kg of body weight, or 1,200 mg in two administrations for those >75 Kg) for 12 weeks.
  Other Names: Rebetol

SUMMARY:
In this pilot study, the investigators plan to treat patients with chronic hepatitis C due to HCV genotype 3 infection using an interferon-free regimen consisting in the administration of ribavirin and sofosbuvir/ledipasvir - a combination of a nucleotide RNA polymerase inhibitor with a non-structural protein 5A inhibitor. Patients will undergo a euglycemic hyperinsulinemic clamp, using tracers, and indirect calorimetry to assess whether the viral suppression induced by this regimen will be capable of reversing the glucose metabolic alterations induced by HCV in both the liver and extrahepatic compartments. Adipose and muscle tissue biopsies will also be performed to assess some specific molecular changes induced by HCV.

DETAILED DESCRIPTION:
Epidemiological studies have shown that hepatitis C virus (HCV) infection induces insulin resistance, which may progress to type 2 diabetes in susceptible individuals. Despite the fact that HCV infects the liver, insulin resistance in these patients appears to originate mostly in extrahepatic tissues, particularly in muscles and adipose tissues. The aim of this trial is to assess the relative contribution of hepatic vs. extrahepatic tissues to the pathogenesis of insulin resistance in chronic hepatitis C. To do so, 20 patients will be enrolled in a single-arm, open-label study. Study subjects will include 10 patients without any feature of the metabolic syndrome, and another 10 with the metabolic syndrome. All patients will receive the same regimen consisting of Ledipasvir 90 mg/Sofosbuvir 400 mg, one tablet once a day, associated with body weight-dose adjusted, 200 mg-tablets of ribavirin (1,000 mg in two administration in patients <75 Kg of body weight, or 1,200 mg in two administrations for those >75 Kg) for 12 weeks. Insulin resistance will be investigated at baseline (before treatment) and after 6 weeks of treatment using a euglycemic hyperinsulinemic clamp with deuterated glucose: results obtained at 6 weeks - i.e. at the time of complete viral suppression - will be compared to basal conditions i.e. before antiviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic hepatitis C with HCV genotype 3a infection,
* Adult Caucasian patient males or non-pregnant or non-lactating females, aged 18 to 65 at the time of the screening;
* Informed Consent as documented by signature;
* Lack of contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational products.

Exclusion Criteria:

* Cirrhosis;
* Excess active alcohol consumption (>30 g/day in males, >20 g/day in females);
* Active illicit drug use.
* Coinfection with HIV or hepatitis B virus;
* Concomitant medications with clinically significant interactions with the study drugs;
* Women who are pregnant or breast feeding or who intend to become pregnant during the course of the study;
* Lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases;
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.);
* Known or suspected non-compliance;
* Inability to follow the procedures of the study, including, but not limited to, language problems, psychological disorders, dementia;
* Participation in another study with any investigational drug within the 30 days preceding and during the present study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Hepatitis C virus-induced insulin resistance | 6 weeks
  Increased (equal to or higher than 10% vs. basal) glucose consumption in patients with chronic hepatitis C but without the metabolic syndrome after complete suppression of viral replication induced by 6 weeks of treatment with Ledipasvir 90 mg/Sofosbuvir 400 mg and ribavirin, as measured by euglycemic hyperinsulinemic clamp using deuterated glucose, and compared to basal conditions i.e. before antiviral treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Negro, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Division of Gastroenterology and hepatology, University Hospital, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Scientific publication in a peer-reviewed journal